CLINICAL TRIAL: NCT05398484
Title: A Phase 2b, Randomized, Double-blind, Placebo-controlled, Multi-center Study of the Effects of Psilocybin-assisted Psychotherapy on Psychiatric and Existential Distress in Advanced Cancer
Brief Title: Psilocybin Therapy in Advanced Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-00498
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Niacin; Psychotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants receiving Study Drug (Experimental): Advanced cancer participants will receive experimental medication, psilocybin (25mg). In addition to the pharmacologic intervention, participants will receive a manualized psychotherapy platform. The combination of interventions is referred to as psilocybin-assisted psychotherapy (PAP).
  Interventions: Drug: Psilocybin 25 mgs; Behavioral: Psychotherapy
- Participants receiving Placebo (Active Comparator): Advanced cancer participants will receive active placebo - single dose of niacin (100mg). In addition to the placebo, participants will receive the same manualized psychotherapy platform as the experimental arm.
  Interventions: Drug: Niacin 100mg; Behavioral: Psychotherapy

INTERVENTIONS:
Drug: Psilocybin 25 mgs — One capsule containing 25mg of psilocybin will be administered with water orally. The appearance of psilocybin is Size 2 HPMC opaque.
  Arms: Participants receiving Study Drug
Drug: Niacin 100mg — One capsule contains 100mg of niacin will be administered with water orally. The appearance of the active placebo is Size 2 HPMC opaque.
  Arms: Participants receiving Placebo
Behavioral: Psychotherapy — The manualized psychotherapy platform will consist of 6 hours of preparatory psychotherapy (prior to the single medication session) and 8 hours of integration psychotherapy following the dosing session.

SUMMARY:
The purpose of this research is to study the safety and effects of single-dose psilocybin 25mg versus an active placebo (single dose niacin 100mg) in the treatment of anxiety, depression, and existential distress (i.e., loss of meaning and hope; fear of death) in advanced cancer (i.e., stage 3 or 4). Study medications will be administered in conjunction with brief psychotherapy that is designed to treat anxiety, depression and existential distress in advanced cancer.

DETAILED DESCRIPTION:
This trial is designed to evaluate efficacy and psychological mechanisms of single-dose psilocybin-assisted psychotherapy (PAP) to treat psychiatric (anxiety, depression) and existential distress (demoralization, death anxiety), and quality-of-life (QOL), in 200 outpatients with late-stage or advanced cancer. The study will assess the strength and durability of therapeutic effects in a double-blind, parallel-design, placebo-controlled, two-center RCT comparing a single 25mg oral 'high' dose of psilocybin to a single 100mg dose of niacin (active placebo), both delivered in conjunction with a psychotherapy platform.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 21
* Diagnosis of Advanced Cancer defined as:

  * Solid tumors to include stage 3 or 4, metastatic illness, or recurrent illness
  * Hematologic malignancies to include, but not limited to, Stage 3 or 4 non-Hodgkins lymphoma, late-stage multiple myeloma or second-line therapy for multiple myeloma, and all forms of acute myeloid leukemia
* Functional Status defined as: Eastern Cooperative Oncology Group (ECOG) ≤2 and Palliative Performance Scale (PPS) ≥60%
* Clinically significant Anxiety defined as SIGH-A >17 at Screening
* Have an identified support person: agree to be accompanied home (or to an otherwise safe destination) by the support person, or another responsible party, following dosing
* Participants of childbearing potential must agree to practice an effective means of birth control throughout the duration of the study. A person of childbearing potential is anyone assigned female or intersex at birth who has experienced menarche and who has not undergone surgical sterilization (e.g., hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or has not completed menopause. Menopause is defined clinically as 12 months of amenorrhea in a person over age 45 in the absence of other biological, physiological, or pharmacological causes.

Exclusion Criteria:

* Unstable medical conditions or serious abnormalities of complete blood count, chemistries, or ECG that in the opinion of the study physician would preclude safe participation in the trial. Some examples include:

  * Congestive heart failure
  * Clinically significant arrhythmias (e.g., ventricular fibrillation, torsades) or clinically significant ECG abnormality (i.e., QTC interval > 450)
  * Recent acute myocardial infarction or evidence of ischemia
  * Malignant hypertension
  * Congenital long QT syndrome
  * Acute renal failure
  * Severe hepatic impairment
  * Respiratory failure
* Risk for hypertensive crisis defined as Screening, Baseline, and Medication Session (prior to dosing) Blood Pressure >140/90 mmHg.
* Significant central nervous system (CNS) pathology. Some examples include:

  * Primary or secondary cerebral neoplasm
  * Epilepsy
  * History of stroke
  * Cerebral aneurysm
  * Dementia
  * Delirium
* Primary psychotic or affective psychotic disorders. Some examples include current or past DSM-5 criteria for:

  * Schizophrenia spectrum disorders
  * Schizoaffective disorder
  * Bipolar I with psychotic features
  * Major Depressive Disorder with psychotic features
* Family history of first-degree relative with psychotic or serious bipolar spectrum illness. Examples include first-degree relative with:

  * Schizophrenia spectrum disorders
  * Schizoaffective disorder
  * Bipolar I with psychotic features
* High risk of adverse emotional or behavioral reaction based on investigator's clinical evaluation. Examples include:

  * Agitation
  * Violent behavior
* Active substance use disorders (SUDs) defined as: DSM-5 criteria for alcohol or drug use disorder (excluding caffeine and nicotine) within the past year
* Extensive use of serotonergic hallucinogens (e.g., LSD, psilocybin) defined as:

  * Any use in the last 12 months
  * >25 lifetime uses
* Clinically significant suicidality or high risk of completed suicide defined as:

  * Active suicidal behavior (interrupted or aborted attempt; preparatory acts) as assessed by Baseline Version of C-SSRS. If C-SSRS items are 4 or 5, participant is ineligible
  * History of suicide attempt(s) within the past year
  * Have any suicidal ideation or thoughts, in the opinion of the study physician or PI, that presents a serious risk of suicidal or self-injurious behavior
* History of hallucinogen persisting perception disorder (HPPD)
* Cognitive impairment as defined by: Montreal Cognitive Assessment Test (MoCA) < 23
* Concurrent Medications

  * Antidepressants
  * Centrally-acting serotonergic agents (e.g., MAO inhibitors)
  * Antipsychotics (e.g., first and second generation)
  * Mood stabilizers (e.g., lithium, valproic acid)
  * Aldehyde dehydrogenase inhibitors (e.g., disulfiram)
  * Significant inhibitors of UGT 1A0 or UGT 1A10
  * Niacin. Note: If taking any supplement containing niacin, agrees to suspend use for at least five days prior to dosing and for the duration of the study
* Have a positive urine drug test including Amphetamines, Barbiturates, Buprenorphine, Benzodiazepines, Cocaine, Cannabis, Methamphetamine, MDMA, Methadone, Opiates (Morphine, Oxycodone), Phencyclidine (PCP), and Tetrahydrocannabinol (THC).

  * Note: Prescribed opiate medications (e.g., cancer-related pain) will be allowed to continue through the study period for participants who have been on a stable dose of such medicine for at least 1 month prior to Screening, as determined during review of concomitant medications.
  * Note: Prescribed benzodiazepine medications and non-benzodiazepine sleeping medications will be allowed to continue through the study period for participants who have been on a stable dose of such a medicine for at least 6 weeks prior to Screening, as determined during review of concomitant medications.
  * Note: Participants using cannabis, including legal cannabis, for any purposes must agree to refrain from use beginning at Screening, as confirmed with a negative Baseline drug test, and through to the end of the study.
  * Note: Participants using prescribed psychostimulants (amphetamines and Ritalin), must agree to refrain from use two weeks prior to baseline visit, as confirmed with a negative Baseline drug test, and through to the end of the study.
* Have a psychiatric condition judged to be incompatible with establishment of rapport with the study therapists or safe exposure to psilocybin
* Participants who are pregnant, as indicated by a positive urine pregnancy test at Screening, Baseline, or prior to dosing on medication administration sessions. Participants who intend to become pregnant during the study or who are currently nursing.
* Have any psychological or physical symptom, medication or other relevant finding prior to randomization, based on the clinical judgment of the PI or relevant clinical study staff that would make a participant unsuitable for the study.
* Have an allergy or intolerance to any of the materials contained in either drug product
* Be enrolled in another clinical trial assessing intervention(s) for anxiety, depression, and/or existential distress (e.g., pharmacologic or psychotherapeutic interventions)

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Structured Interview Guide for the Hamilton Anxiety Scale (HAM-A): SIGH-A Score | Baseline, Week 8
  Structured Interview Guide for the Hamilton Anxiety Scale (SIGH-A) measures the level of anxiety in participants. Scoring is based on a 17-item scale and scores of 0-7 are considered as being normal, 8-16 suggest mild anxiety, 17-23 moderate anxiety, and scores over 24 are indicative of severe anxiety; the maximum score being 52.

SECONDARY OUTCOMES:
Change in Structured Interview Guide for the Montgomery-Asberg Depression Rating Scale (MADRS): SIGMA Score | Baseline, Week 8
  Structured Interview Guide for the Montgomery-Asberg Depression Rating Scale (SIGMA) measures the level of depression in participants. Scoring is based on a 10-item rating scale and each item is rated on a 0 (least severe) to 6 (most severe) scale, resulting in a maximum total score of 60 points.
Change in Structured Interview Guide for the Montgomery-Asberg Depression Rating Scale (MADRS): SIGMA Score | Baseline, Week 12
  Structured Interview Guide for the Montgomery-Asberg Depression Rating Scale (SIGMA) measures the level of depression in participants. Scoring is based on a 10-item rating scale and each item is rated on a 0 (least severe) to 6 (most severe) scale, resulting in a maximum total score of 60 points.
Change in Structured Interview Guide for the Montgomery-Asberg Depression Rating Scale (MADRS): SIGMA Score | Baseline, Month 6
  Structured Interview Guide for the Montgomery-Asberg Depression Rating Scale (SIGMA) measures the level of depression in participants. Scoring is based on a 10-item rating scale and each item is rated on a 0 (least severe) to 6 (most severe) scale, resulting in a maximum total score of 60 points.
Change in Hospital Anxiety and Depression Scale (HADS) - Depression Subscale Score | Baseline, Week 8
  The Hospital Anxiety and Depression Scale (HADS) comprises seven questions about depression. The total score range is 0-21 with each answer ranging from 0 (absence) to 3 (extreme presence). Higher scores indicate greater levels of depression.
Change in Hospital Anxiety and Depression Scale (HADS) - Depression Subscale Score | Baseline, Week 12
  The Hospital Anxiety and Depression Scale (HADS) comprises seven questions about depression. The total score range is 0-21 with each answer ranging from 0 (absence) to 3 (extreme presence). Higher scores indicate greater levels of depression.
Change in Hospital Anxiety and Depression Scale (HADS) - Depression Subscale Score | Baseline, Month 6
  The Hospital Anxiety and Depression Scale (HADS) comprises seven questions about depression. The total score range is 0-21 with each answer ranging from 0 (absence) to 3 (extreme presence). Higher scores indicate greater levels of depression.
Change in Hospital Anxiety and Depression Scale (HADS) - Anxiety Subscale Score | Baseline, Week 8
  The Hospital Anxiety and Depression Scale (HADS) comprises seven questions about anxiety. The total score range is 0-21 with each answer ranging from 0 (absence) to 3 (extreme presence). Higher scores indicate greater levels of anxiety.
Change in Hospital Anxiety and Depression Scale (HADS) - Anxiety Subscale Score | Baseline, Week 12
  The Hospital Anxiety and Depression Scale (HADS) comprises seven questions about anxiety. The total score range is 0-21 with each answer ranging from 0 (absence) to 3 (extreme presence). Higher scores indicate greater levels of anxiety.
Change in Hospital Anxiety and Depression Scale (HADS) - Anxiety Subscale Score | Baseline, Month 6
  The Hospital Anxiety and Depression Scale (HADS) comprises seven questions about anxiety. The total score range is 0-21 with each answer ranging from 0 (absence) to 3 (extreme presence). Higher scores indicate greater levels of anxiety.
Changes in Demoralization Scale Version II (DS-II) Score | Baseline, Week 8
  The Demoralization Scale Version II (DS-II) is a validated and frequently used instrument to assess existential distress in patients with cancer and other severe medical illness. Items are rated on a 3-point Likert scale ranging from 0 (never) to 2 (often), with two subscales (Meaning and Purpose; Distress & Coping Ability). A total score for demoralization is calculated by summarizing the single subscale scores; the total score range is 0-32. Higher scores indicate higher levels of demoralization.
Changes in Demoralization Scale Version II (DS-II) Score | Baseline, Week 12
  The Demoralization Scale Version II (DS-II) is a validated and frequently used instrument to assess existential distress in patients with cancer and other severe medical illness. Items are rated on a 3-point Likert scale ranging from 0 (never) to 2 (often), with two subscales (Meaning and Purpose; Distress & Coping Ability). A total score for demoralization is calculated by summarizing the single subscale scores; the total score range is 0-32. Higher scores indicate higher levels of demoralization.
Changes in Demoralization Scale Version II (DS-II) Score | Baseline, Month 6
  The Demoralization Scale Version II (DS-II) is a validated and frequently used instrument to assess existential distress in patients with cancer and other severe medical illness. Items are rated on a 3-point Likert scale ranging from 0 (never) to 2 (often), with two subscales (Meaning and Purpose; Distress & Coping Ability). A total score for demoralization is calculated by summarizing the single subscale scores; the total score range is 0-32. Higher scores indicate higher levels of demoralization.
Change in Death and Dying Distress Scale Version 2 (DADDS-2) Score | Baseline, Week 8
  Death and Dying Distress Scale Version 2 (DADDS-2) scale is a 15-item self-report measure assessing distress regarding awareness of shortness of time and the process of dying, specifically in patients with advanced cancer. The total score range is 0-75. Higher Scores indicate greater death distress.
Change in Death and Dying Distress Scale Version 2 (DADDS-2) Score | Baseline, Week 12
  Death and Dying Distress Scale Version 2 (DADDS-2) scale is a 15-item self-report measure assessing distress regarding awareness of shortness of time and the process of dying, specifically in patients with advanced cancer. The total score range is 0-75. Higher Scores indicate greater death distress.
Change in Death and Dying Distress Scale Version 2 (DADDS-2) Score | Baseline, Month 6
  Death and Dying Distress Scale Version 2 (DADDS-2) scale is a 15-item self-report measure assessing distress regarding awareness of shortness of time and the process of dying, specifically in patients with advanced cancer. The total score range is 0-75. Higher Scores indicate greater death distress.
Change in Death Transcendence Scale (DTS) Score | Baseline, Week 8
  Death Transcendence Scale (DTS) is a 15-item self-report measure assessing distress regarding awareness of shortness of time and the process of dying, specifically in patients with advanced cancer. The total score range is 0-75. Higher Scores indicate greater death distress.
Change in Death Transcendence Scale (DTS) Score | Baseline, Week 12
  Death Transcendence Scale (DTS) is a 15-item self-report measure assessing distress regarding awareness of shortness of time and the process of dying, specifically in patients with advanced cancer. The total score range is 0-75. Higher Scores indicate greater death distress.
Change in Death Transcendence Scale (DTS) Score | Baseline, Month 6
  Death Transcendence Scale (DTS) is a 15-item self-report measure assessing distress regarding awareness of shortness of time and the process of dying, specifically in patients with advanced cancer. The total score range is 0-75. Higher Scores indicate greater death distress.
Change in Functional Assessment of Cancer Therapy-General (FACT-G) Score | Baseline, Week 8
  The Functional Assessment of Cancer Therapy - General (FACT-G) is a 27-item questionnaire designed to measure four domains of Health-related quality of life (HRQOL) in cancer patients: Physical, social, emotional, and functional well-being. All questions in the FACT-G use a 5-point rating scale (0 = Not at all; 1 = A little bit; 2 = Somewhat; 3 = Quite a bit; and 4 = Very much). The FACT-G total score is computed as the sum of the four subscale scores, provided the overall item response is at least 80% (i.e., at least 22 of the 27 items were answered) and has a possible range of 0-108 points. The lower the score, the greater the quality of life
Change in Functional Assessment of Cancer Therapy-General (FACT-G) Score | Baseline, Week 12
  The Functional Assessment of Cancer Therapy - General (FACT-G) is a 27-item questionnaire designed to measure four domains of Health-related quality of life (HRQOL) in cancer patients: Physical, social, emotional, and functional well-being. All questions in the FACT-G use a 5-point rating scale (0 = Not at all; 1 = A little bit; 2 = Somewhat; 3 = Quite a bit; and 4 = Very much). The FACT-G total score is computed as the sum of the four subscale scores, provided the overall item response is at least 80% (i.e., at least 22 of the 27 items were answered) and has a possible range of 0-108 points. The lower the score, the greater the quality of life
Change in Functional Assessment of Cancer Therapy-General (FACT-G) Score | Baseline, Month 6
  The Functional Assessment of Cancer Therapy - General (FACT-G) is a 27-item questionnaire designed to measure four domains of Health-related quality of life (HRQOL) in cancer patients: Physical, social, emotional, and functional well-being. All questions in the FACT-G use a 5-point rating scale (0 = Not at all; 1 = A little bit; 2 = Somewhat; 3 = Quite a bit; and 4 = Very much). The FACT-G total score is computed as the sum of the four subscale scores, provided the overall item response is at least 80% (i.e., at least 22 of the 27 items were answered) and has a possible range of 0-108 points. The lower the score, the greater the quality of life
Change in Functional Assessment of Chronic Illness Therapy-Spiritual well-being, 12-items (FACIT-Sp-12) Score | Baseline, Week 8
  The Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being (FACIT-Sp-12) is a 12-item questionnaire that measures spiritual well-being in people with cancer and other chronic illnesses. Answers are scored on a 5-point Likert scale from 0 to 4. Total scores range from 0 to 48, higher scores indicating higher spiritual well-being.
Change in Functional Assessment of Chronic Illness Therapy-Spiritual well-being, 12-items (FACIT-Sp-12) Score | Baseline, Week 12
  The Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being (FACIT-Sp-12) is a 12-item questionnaire that measures spiritual well-being in people with cancer and other chronic illnesses. Answers are scored on a 5-point Likert scale from 0 to 4. Total scores range from 0 to 48, higher scores indicating higher spiritual well-being.
Change in Functional Assessment of Chronic Illness Therapy-Spiritual well-being, 12-items (FACIT-Sp-12) Score | Baseline, Month 6
  The Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being (FACIT-Sp-12) is a 12-item questionnaire that measures spiritual well-being in people with cancer and other chronic illnesses. Answers are scored on a 5-point Likert scale from 0 to 4. Total scores range from 0 to 48, higher scores indicating higher spiritual well-being.
Change in Clinical Global Impression - Severity of Illness (CGI-S) Score | Baseline, Week 8
  Clinical Global Impression - Severity of Illness (CGI-S) is a standardized assessment scale for determining the effects of mental health treatment among patients with psychiatric illnesses and measures symptom severity, intervention response and the efficacy of interventions in intervention studies of patients with mental disorders. It is a 7-item clinician-administered questionnaire scoring severity of current illness from Normal, not ill at all (1) to Among the most extremely ill patients (7).
Change in Clinical Global Impression - Severity of Illness (CGI-S) Score | Baseline, Week 12
  Clinical Global Impression - Severity of Illness (CGI-S) is a standardized assessment scale for determining the effects of mental health treatment among patients with psychiatric illnesses and measures symptom severity, intervention response and the efficacy of interventions in intervention studies of patients with mental disorders. It is a 7-item clinician-administered questionnaire scoring severity of current illness from Normal, not ill at all (1) to Among the most extremely ill patients (7).
Change in Clinical Global Impression - Severity of Illness (CGI-S) Score | Baseline, Month 6
  Clinical Global Impression - Severity of Illness (CGI-S) is a standardized assessment scale for determining the effects of mental health treatment among patients with psychiatric illnesses and measures symptom severity, intervention response and the efficacy of interventions in intervention studies of patients with mental disorders. It is a 7-item clinician-administered questionnaire scoring severity of current illness from Normal, not ill at all (1) to Among the most extremely ill patients (7).
Change in Clinical Global Impression - Improvement (CGI-I) Score | Baseline, Week 8
  Clinical Global Impression - Improvement (CGI-I) is a standardized assessment scale for rating a participant's global improvement relative to treatment intervention. It is a 7-item clinician-administered questionnaire scoring improvement of current illness from Much Improved (1) to Very much Worse (7).
Change in Clinical Global Impression - Improvement (CGI-I) Score | Baseline, Week 12
  Clinical Global Impression - Improvement (CGI-I) is a standardized assessment scale for rating a participant's global improvement relative to treatment intervention. It is a 7-item clinician-administered questionnaire scoring improvement of current illness from Much Improved (1) to Very much Worse (7).
Change in Clinical Global Impression - Improvement (CGI-I) Score | Baseline, Month 6
  Clinical Global Impression - Improvement (CGI-I) is a standardized assessment scale for rating a participant's global improvement relative to treatment intervention. It is a 7-item clinician-administered questionnaire scoring improvement of current illness from Much Improved (1) to Very much Worse (7).
Change in Persisting Effects Questionnaire (PEQ) Score | Week 8, Month 6
  Persisting Effects Questionnaire (PEQ) Score is a self-report measure that was designed to assess positive and negative changes in moods, attitudes, behavior, as well as meaningfulness and spiritual significance attributed to psilocybin administration. The abbreviated questionnaire has 14 items pertaining to the participant's experience as it relates to various aspects of life and whether it has led to long-term and persisting changes.
Mystical Experience Questionnaire-30 items (MEQ-30) Score | 8 hours post-medication
  The Mystical Experience Questionnaire (MEQ) is an unvalidated self-report measure that has been used to measure mystical-type experiences in laboratory studies of hallucinogens. Scoring consists of 0 - none; not at all; 1 - so slight cannot decide; 2 - slight; 3- moderate; 4 - strong (equivalent in degree to any other strong experience); 5- extreme (more than any other time in my life and stronger than 4). MEQ30 total scores range from 0 to 150; the higher the score, the greater the mystical-type experiences occasioned by psilocybin

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ross, MD, Principal Investigator — NYU Langone Medical Center
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical campus (CU AMC), Aurora, Colorado
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request. Requests should be directed to Stephen.ross@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Schipper S, Nigam K, Schmid Y, Piechotta V, Ljuslin M, Beaussant Y, Schwarzer G, Boehlke C. Psychedelic-assisted therapy for treating anxiety, depression, and existential distress in people with life-threatening diseases. Cochrane Database Syst Rev. 2024 Sep 12;9(9):CD015383. doi: 10.1002/14651858.CD015383.pub2. PMID 39260823